CLINICAL TRIAL: NCT06682949
Title: Daily Routines and Executive Functioning in Youth with ADHD
Brief Title: Daily Routines, Executive Functioning & ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cori Manning (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor-Investigator, Cori Manning, Doctoral Candidate of School Psychology, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003784
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Attention Deficit Disorder with Hyperactivity (ADHD)
Keywords: ADHD; executive function; attention; adolescent; working memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Extension (Experimental): Participants will review their baseline actigraphy data with a research team member and discuss sleep patterns. Participants will be given a "sleep prescription", giving them specified sleep and wake times based on AASM guidelines. Participants and their parent will discuss stimulus control with team member. Participants will implement their sleep prescription for two weeks.
  Interventions: Behavioral: Sleep Extension
- Daytime Routine (Placebo Comparator): Participants will review their daily routines with a research team member. With parent collaboration, they will agree to adjust a behavioral daytime routine to implement for the next two weeks.
  Interventions: Behavioral: Daytime Routine

INTERVENTIONS:
Behavioral: Sleep Extension — Participants, their parent, and a researcher will review the participants actigraphy data from the two week baseline period. They will discuss sleep patterns and behaviors related to sleep. The researcher will prescribe a sleep prescription that includes set sleep and wake times and stimulus control. Participants will adhere to the sleep prescription for two weeks.
  Arms: Sleep Extension
Behavioral: Daytime Routine — Participant, their parent, and researcher will meet to discuss daily routines for the child and family. They will collaborate to choose one behavioral routine to modify for the following two weeks.
  Arms: Daytime Routine

SUMMARY:
The goal of this clinical trial is to learn adjusting daily or nightly routines improves executive functioning in youth with ADHD. It will also learn about the acceptability of the intervention.

The main questions it aims to answer are:

1. Does the intervention improve sleep for youth with ADHD?
2. Does the intervention improve areas of executive functioning for youth with ADHD?
3. Is this an acceptable intervention for youth with ADHD?

Researchers will compare the two intervention conditions to see if their are impacts in executive functioning and sleep.

Participants will:

Complete cognitive testing, executive function tasks, questionnaires, and an interview at baseline and at one month Wear an actigraph watch for one month Bring a parent with them to three meetings Complete daily sleep diaries for one month

DETAILED DESCRIPTION:
The purpose of this study will be to examine if adolescents with ADHD with altered daily or nightly routines show improvements in EF, specifically working memory, cognitive flexibility, and inhibitory control. This will be a pilot study including up to 25 adolescents between the ages of 11 and 17 years old, with a diagnosis of ADHD (combined presentation, or predominantly inattentive presentation). Participants will be stratified by gender and randomly assigned to one of two conditions: 1) night routines or 2) daily routines. The intervention is ready to be implemented and adapted for an ADHD population. Though the intervention itself was not focused on sleep hygiene, the team incorporated strategies to increase the likelihood of extending sleep duration, such as reviewing actigraphy and sleep diary data with the participant, collaboration between the participant, caregiver and researcher to address obstacles to obtaining enough sleep, and instructing the participant to obtain a specific amount of sleep. The first study demonstrated that sleep extension in youth with type 1 diabetes (T1DM) was feasible, whereas the ongoing study has demonstrated that overall youth increase TST over a 3-month period. This latter study has a booster session approximately one month after the initial consultation. Thus, this study will last one month with two weeks of baseline to establish sleep patterns and the intervention portion for this study will last for two weeks to monitor whether the youth increase their sleep and ascertain an effect size of intervention impact.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of attention-deficit/hyperactivity disorder (ADHD)
* Located in the greater Tucson, AZ area
* Must have a guardian willing to participate

Exclusion Criteria:

* Clinical diagnosis of autism spectrum disorder
* Clinical diagnosis of an intellectual disability
* Clinical diagnosis of psychosis
* Clinical diagnosis of bipolar disorder

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sleep duration | Beginning at consent meeting and lasting four weeks
  Actigraphy data will be used to determine changes in sleep duration pre and post intervention. Average total sleep time during the baseline period will be compared to average total sleep time during the intervention period.
Sleep Consistency | Beginning at consent meeting (day 1) and ending at final meeting (day 28)
  Actigraphy data will be used to determine changes in consistency of sleep periods. Average sleep periods will be compared pre and post intervention.
Sleep Quality | Begin day 1 and end day 28
  The Children's Report of Sleep Patterns will be completed at baseline and post intervention to evaluate any changes in reported overall sleep quality.

SECONDARY OUTCOMES:
Executive Functioning - Working Memory | From consent to the one month mark
  Participants will complete a computerized version Digit Span (backward) at baseline and at the post intervention meeting. Pre and post scores will be compared to determine change in working memory. Higher scores of longest digit span recalled indicate better auditory working memory. Min = 0, Max = 9
Executive Functioning - Cognitive Flexibility (set-shifting) | Begin at day 1 and end at day 28
  Participants will complete a digital version of the trail making task at baseline and post intervention. Scores at pre and post will be compared to evaluate any change in cognitive flexibility, also know as set-shifting. Total errors and total time for completion are measured. Higher scores on both indicate wose cognitive flexibility
Executive functioning - Inhibitory control | Begin day 1 and end day 28
  Participants will complete a digital version of the stop signal task at baseline and at the post intervention meeting. Scores will be compared to evaluate any change in inhibitory control. Z scores are calculated to compare abilities to a normative sample. Scores range from -3 to 3 with negative scores reflecting worse performance.
General Executive Functioning | Begin day 1 and end day 28
  The BRIEF will be completed pre and post intervention as a subjective measure of executive functioning as a whole. Scores will be compared at pre and post to evaluate any change index scores. T-scores are produced with scores at or above 65 indicate clinical significance.

OTHER OUTCOMES:
Acceptibility of the intervention among youth with ADHD | At the four week mark.
  At the final meeting (week 4), participants will participate in an acceptability interview to determine if the intervention is acceptable within this population.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Perfect, PhD, Study Chair — University of Arizona
Locations (1):
- University of Arizona - College of Education, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perfect MM, Silva GE, Chin CN, Wheeler MD, Frye SS, Mullins V, Quan SF. Extending sleep to improve glycemia: The Family Routines Enhancing Adolescent Diabetes by Optimizing Management (FREADOM) randomized clinical trial protocol. Contemp Clin Trials. 2023 Jan;124:106929. doi: 10.1016/j.cct.2022.106929. Epub 2022 Sep 19. PMID 36441106
- [Background] Perfect MM, Beebe D, Levine-Donnerstein D, Frye SS, Bluez GP, Quan SF. The Development of a Clinically Relevant Sleep Modification Protocol for Youth with Type 1 Diabetes. Clin Pract Pediatr Psychol. 2016 Jun;4(2):227-240. doi: 10.1037/cpp0000145. PMID 27747146
- [Background] Becker SP, Duraccio KM, Sidol CA, Fershtman CEM, Byars KC, Harvey AG. Impact of a Behavioral Sleep Intervention in Adolescents With ADHD: Feasibility, Acceptability, and Preliminary Effectiveness From a Pilot Open Trial. J Atten Disord. 2022 May;26(7):1051-1066. doi: 10.1177/10870547211056965. Epub 2021 Nov 5. PMID 34738484
- [Background] Larsson I, Aili K, Lonn M, Svedberg P, Nygren JM, Ivarsson A, Johansson P. Sleep interventions for children with attention deficit hyperactivity disorder (ADHD): A systematic literature review. Sleep Med. 2023 Feb;102:64-75. doi: 10.1016/j.sleep.2022.12.021. Epub 2022 Dec 26. PMID 36603513
- [Background] Malkani MK, Pestell CF, Sheridan AMC, Crichton AJ, Horsburgh GC, Bucks RS. Behavioral Sleep Interventions for Children With ADHD: A Systematic Review and Meta-Analysis. J Atten Disord. 2022 Dec;26(14):1805-1821. doi: 10.1177/10870547221106239. Epub 2022 Jun 25. PMID 35758199